CLINICAL TRIAL: NCT02464540
Title: Randomized Clinical Trial of Light Cured Luting Agents on Laminate Veneers
Brief Title: Optical Properties of Light Cured Luting Agent on Laminate Veneer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Noéli Boscato, PhD, Adjunct Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUPelotas
Record Dates: First submitted 2015-05-08; First posted 2015-06-08 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Optical Properties of Laminate Veneers
Keywords: laminate veneers; luting agent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Light-cured resin cement (Active Comparator): Laminate veneers luted using light-cured resin cement
  Interventions: Procedure: Laminate veneers luted with light-cured resin cement
- Light-cured flowable composite (Active Comparator): Laminate veneers luted using light-cured flowable composite
  Interventions: Procedure: Laminate veneers luted with light-cured flowable composite

INTERVENTIONS:
Procedure: Laminate veneers luted with light-cured resin cement — After the use of light-cured luting agent the color of laminate venners will be performed with visual evaluation based on Vita and 3D Master scales and with a spectrophotometer Vita Easyshade (Vita Zahnfabrik / Bad Saeckingen, Germany) based on CIEL*a* b system. Data collected will be evaluated for translucency parameter (TP) and color variation (ΔE) according to luting agent, thickness and color of the LVs as well as color of dental substrate. Additionally, the color obtained with visual evaluation and with spectrophotometer will be compared to evaluate the level of agreement between the color observed by the operator and the color named by the spectrophotometer.
  Arms: Light-cured resin cement
Procedure: Laminate veneers luted with light-cured flowable composite — After the use of light-cured luting agent the color of laminate veneers will be performed with visual evaluation based on Vita and 3D Master scales and with a spectrophotometer Vita Easyshade (Vita Zahnfabrik / Bad Saeckingen, Germany) based on CIEL*a* b system. Data collected will be evaluated for translucency parameter (TP) and color variation (ΔE) according to luting agent, thickness and color of the LVs as well as color of dental substrate. Additionally, the color obtained with visual evaluation and with spectrophotometer will be compared to evaluate the level of agreement between the color observed by the operator and the color named by the spectrophotometer.
  Arms: Light-cured flowable composite

SUMMARY:
The aim of this randomized clinical trial is to evaluate the influence of luting agent, thickness and color of laminate veneers (LVs) and color of dental substrate on the optical properties of LVs.

DETAILED DESCRIPTION:
The following date will be collected (i) the color of dental substrate obtained before and after dental preparation, (ii) the thickness and color of the LVs obtained before of the cementation procedures on white and black value background, (iii) and the final color of the LVs bonded to dental substrates obtained after cementation. For LVs cementation two cements will be used, the light-cured resin cement and the flowable composite, which will be randomly divided into two groups (n=31). The color of LVs will be performed with visual evaluation based on Vita and 3D Master scales and with a spectrophotometer Vita Easyshade (Vita Zahnfabrik / Bad Saeckingen, Germany) based on CIEL*a* b system. Data collected will be evaluated for translucency parameter (TP) and color variation (ΔE) according to luting agent, thickness and color of the LVs as well as color of dental substrate. Additionally, the color obtained with visual evaluation and with spectrophotometer will be compared to evaluate the level of agreement between the color observed by the operator and the color named by the spectrophotometer.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Patients with diastema
* Conoid teeth
* Misaligned anterior teeth
* Discolored teeth and/or teeth with erosion/abrasion
* Posterior occlusal stability
* Individuals who are willing to attend the clinics on predetermined days, to agree to sign the consent form and clarified, after receiving information about the study objectives, risks and benefits associated with the procedures.

Exclusion Criteria:

* Patients with extensive loss of tooth structure
* Subjects suffering from temporomandibular disorders, neurological and oral mucosa diseases
* Inadequate oral hygiene or periodontal problems
* Smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noéli Boscato, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Noéli Boscato, Pelotas, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: ceramic restoration
Groups:
- Light-cured Resin Cement: Ceramic restorations were cemented using translucent shade of photoactivated resin cement (RelyX Veneer; 3M ESPE).
- Light-cured Flowable Composite: Ceramic restorations were cemented using translucent shade of flowable composite (Tetric N-Flow; Ivoclar Vivadent AG)
Period: Overall Study
Arm/Group | Light-cured Resin Cement | Light-cured Flowable Composite
Started (Participants enrolled in both arms, luting material to be used was randomly selected.) | 11; 17 ceramic restoration | 11; 21 ceramic restoration
Completed | 11; 17 ceramic restoration | 11; 21 ceramic restoration
Not Completed | 0; 0 ceramic restoration | 0; 0 ceramic restoration

BASELINE CHARACTERISTICS:
Population: 17 restorations cemented with light-cured resin cement and 38 cemented with light-cured flowable composite.
Units Other Than Participants: ceramic restoration
Groups:
- Light-cured Resin Cement - Light-cured Flowable Composite: Ceramic restorations were cemented using translucent shade of photoactivated resin cement or Light-cured flowable composite. Participants enrolled in both arms, luting material to be used was randomly selected.
Arm/Group | Light-cured Resin Cement - Light-cured Flowable Composite
Number analyzed (Participants) | 11
Number analyzed (ceramic restoration) | 38
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 39.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Optical Properties of Laminate Veneers
Description: The color of laminate veneers will be performed with a spectrophotometer Vita Easyshade (Vita Zahnfabrik / Bad Saeckingen, Germany) based on Vita and 3D Master scales and on CIEL*a* b system. Data collected will be evaluated for translucency parameter (TP) and color difference (ΔE) according the thickness and color of the laminate veneers as well as color of dental substrate.
  The acceptable threshold color difference for the CIEDE2000 method is 1.8 (Paravina et al, 2015). Greater color variation is desirable when a shade match between darker and lighter adjacent tooth substrates is required and values above the clinical thresholds for acceptability of color differences indicating lower masking ability of the material.
  "Level of Agreement Between the Color Observed by the Operator and the Color Named by the Spectrophotometer" was included as a Primary or Secondary Outcome Measure, but data was not collected.
Time Frame: after luting the laminate veneers (at least 1 hours after cementation)
Population: 38 ceramic restorations were cemented (25 laminate veneers, 13 crowns; 37 in anterior teeth; 1 in posterior tooth).
Measure: Mean (Standard Deviation); unit: Delta E (color change)
Units Other Than Participants: ceramic restoration
Groups:
- Light-cured Resin Cement; Light-cured Flowable Composite: Color change was estimated by calculating the CIEDE2000 formula. Corresponding ΔE00 values for perceptibility and acceptability were 0.8 and 1.8, respectively. (Paravina, 2015)
Arm/Group | Light-cured Resin Cement | Light-cured Flowable Composite
Number analyzed (Participants) | 11 | 11
Number analyzed (ceramic restoration) | 17 | 21
Delta E (color change) | 5.31 (1.80) | 5.07 (2.37)

ADVERSE EVENTS:
Time Frame: immediately after luting restoration (an average 1 hours after cementation)
Description: Side effects of the dental procedures (pain, fracture, debonding) were recorded.
Groups:
- Light-cured Resin Cement: Ceramic restorations were cemented using translucent shade of photoactivated resin cement.
- Light-cured Flowable Composite: Ceramic restorations were cemented using translucent shade of photoactivated flowable composite.
Arm/Group | Light-cured Resin Cement | Light-cured Flowable Composite
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No